CLINICAL TRIAL: NCT02063243
Title: Intralesional Cryotherapy With a Argon Gas Based Device for the Treatment of Keloid and Hypertrophic Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Michiel van Leeuwen, MD, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12/293
Record Dates: First submitted 2014-02-10; First posted 2014-02-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Keloid; Cicatrix; Hypertrophic
Keywords: Keloid, hypertrophic scar
MeSH Terms: conditions — Keloid; Cicatrix; Hypertrophy; Cicatrix, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- keloid or hypertrophic scars (Other): All patient including all skin types with keloid or hypertrophic disease receiving Intralesional Cryotherapy
  Interventions: Procedure: Intralesional cryotherapy

INTERVENTIONS:
Procedure: Intralesional cryotherapy — Intralesional (IL) cryotherapy is a treatment for keloids and hypertrophic scars, in which the scar is frozen from inside with the use of a cryoneedle
  Other Names: Seednet

SUMMARY:
This prospective evaluation studies the effectiveness of Intralesional (IL) cryotherapy with a argon gas based device in treating keloids and hypertrophic scars in population consisting of all Fitzpatrick skin type patients

DETAILED DESCRIPTION:
Intralesional (IL) cryotherapy is a novel treatment for keloids and hypertrophic scars, in which the scar is frozen from inside. Published results are promising, however only Caucasian patient populations have been studied. This prospective evaluation studies the effectiveness of IL cryotherapy in treating keloids and hypertrophic scars in a population consisting of all Fitzpatrick skin type patients.

Multiple devices are available, mostly based on a simple open system. Closed, argon gas based, systems are highly controlled and provide accurate freezing. However, this technique has never been used for IL cryotherapy for the treatment of keloid or hypertrophic scars. All patients with keloid or hypertrophic scars meeting inclusion criteria were treated with a argon based device called Seednet. Scar quality and possible recurrence are assessed pre- and postsurgery (3, 6 and 12 months) with objective devices determine scar color, scar elasticity, scar volume and patient's skin type. In addition, scars are evaluated using the Patient and Observer Scar Assessment Scale.

ELIGIBILITY:
Inclusion Criteria:

* Keloids, defined as excessive scar tissue raised above skin level and proliferating beyond the confines of the original lesion
* Hypertrophic scars1 older than 12 months and insensitive to other treatments. Keloids were distinguished from hypertrophic scars based on the clinical judgment of experienced plastic surgeons and on the age of the scar (>1yr)
* A period between previous treatment and IL cryotherapy covered a minimum of 12 weeks
* Patients with all Fitzpatrick17 skin types
* Patients older than 10 years of age

Exclusion Criteria:

* pregnancy
* diabetes mellitus

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Recurrence | 0-12 months
  Judgment of recurrence, defined as a growing, pruritic, nodular scar

SECONDARY OUTCOMES:
Scar elasticity | 0-12months
  Scar elasticity, measured in two parameters: extension and elasticity

OTHER OUTCOMES:
Scar volume | 0-12months
  Determined by creating a mold of the scar with dental putty

CONTACTS AND LOCATIONS:
Overall Officials: Michiel CE van Leeuwen, MD, Principal Investigator — VUmc
Locations (1):
- VUmc, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] van Leeuwen MC, Bulstra AE, van Leeuwen PA, Niessen FB. A new argon gas-based device for the treatment of keloid scars with the use of intralesional cryotherapy. J Plast Reconstr Aesthet Surg. 2014 Dec;67(12):1703-10. doi: 10.1016/j.bjps.2014.08.046. Epub 2014 Aug 27. PMID 25257046
- See also: Link Text: homepage VU medical center, hospital Amsterdam, the Netherlands — http://www.vumc.nl